CLINICAL TRIAL: NCT02511132
Title: A 2-part Trial Comparing Overall Survival of Patients With Metastatic Ewing's Sarcoma Treated With Vigil Versus Gemcitabine and Docetaxel and to Determine Safety Profile of Vigil in Combination With Irinotecan and Temozolomide.
Brief Title: A Two-part Phase IIb Trial of Vigil (Bi-shRNAfurin and GMCSF Augmented Autologous Tumor Cell Immunotherapy) in Ewing's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL-121
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Results first posted 2022-07-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Ewing's Sarcoma
Keywords: Ewing's Sarcoma Family of Tumors, ESFT, Sarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing; Sarcoma | interventions — FANG vaccine; Temozolomide; Irinotecan; Gemcitabine; Docetaxel

STUDY DESIGN:
Intervention Model Description: Part 1: Participants will be randomized 1:1 to receive Vigil immunotherapy alone or gemcitabine / docetaxel. Part 2 participants will be a single group of subjects to receive Vigil immunotherapy in combination with irinotecan and temozolomide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Vigil Alone (Experimental): Vigil immunotherapy 1.0 x 107 cells/injection; minimum of 4 to a maximum of 12 administrations every 28 days
  Interventions: Biological: Vigil
- Part 1: Gemicitabine and Docetaxel (Active Comparator): Gemcitabine 675 mg/m2 IV at 10 mg/m2/min D1 and Docetaxel 75 mg/m2 IV starting on D8 and given every 21 days.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel
- Part 2: Vigil plus Temozolomide and Irinotecan (Experimental): (i) oral temozolomide 100 mg/m2 daily (Days 1 - 5, total dose 500 mg/m2/cycle), (ii) irinotecan 50 mg/m2 daily (Days 1 - 5, total dose 250mg/m2/cycle), orally or irinotecan 20mg/m2 daily (Days 1 - 5, total dose 100mg/m2/cycle ), intravenously (iii) peg-filgrastim 100μg/kg (Day 6) subcutaneously (optional and may be administered at home), and (iv) Vigil 1.0 x 107 cells/injection, intradermally on Day 15 and every 3 weeks thereafter. One cycle = 21 days.
  Interventions: Biological: Vigil; Drug: Temozolomide; Drug: Irinotecan

INTERVENTIONS:
Biological: Vigil — Vigil 1.0 x 10e7 cells/injection, minimum of 4 to a maximum of 12 administrations.
  Other Names: formerly known as FANG™; bi-shRNAfurin and GMCSF Autologous Tumor Cell Immunotherapy
  Arms: Part 1: Vigil Alone; Part 2: Vigil plus Temozolomide and Irinotecan
Drug: Temozolomide — oral temozolimidetemozolomide 100 mg/m2 daily (Days 1 - 5, total dose 500 mg/m2/cycle)
  Other Names: TEMODAR
  Arms: Part 2: Vigil plus Temozolomide and Irinotecan
Drug: Irinotecan — irinotecan 50 mg/m2 daily (Days 1 - 5, total dose 250mg/m2/cycle), orally or irinotecan 20mg/m2 daily (Days 1 - 5, total dose 100mg/m2/cycle ), intravenously
  Other Names: CAMPTOSAR
  Arms: Part 2: Vigil plus Temozolomide and Irinotecan
Drug: Gemcitabine — 675 mg/m2 IV at a rate of 10 mg/m2/min on Day 1 and Day 8 every 21 days
  Other Names: GEMZAR
  Arms: Part 1: Gemicitabine and Docetaxel
Drug: Docetaxel — 75 mg/m2 IV administered on Day 8 and every 21 days
  Other Names: TAXOTERE
  Arms: Part 1: Gemicitabine and Docetaxel

SUMMARY:
A two-part trial in patients with metastic Ewing's sarcoma. Participants in Part 1 will be randomized to receive either Vigil immunotherapy or gemcitabine and docetaxel with the objective of comparing the overall survival between the two arms. Participants enrolled in Part 2 will receive Vigil immunotherapy in combination of temozolomide and irinotecan with the objective to determine the safety profile of the combination treatment.

DETAILED DESCRIPTION:
Part 1 Methodology:

This is a multicenter, 1:1 randomized Phase IIb study of intradermal autologous Vigil immunotherapy (1.0 x 10e7 cells/injection; minimum of 4 to a maximum of 12 administrations) versus gemcitabine / docetaxel in patients with metastatic Ewing's sarcoma Family of Tumors (ESFT) refractory or intolerant to at least 2 prior lines of chemotherapy. Patients undergoing a standard surgical procedure (e.g., tumor biopsy or palliative resection) may have tumor tissue harvested for manufacture of investigational product. Patients meeting eligibility criteria including manufacture of a minimum of 4 immunotherapy doses will be randomized to receive either (1) intradermal Vigil every 28 days for 4-12 administrations, or (2) gemcitabine 675 mg/m2 IV at 10 mg/m2/min D1 and D8 and docetaxel 75 mg/m2 IV D8 every 21 days. The primary trial objective is to determine the overall survival of patients treated with Vigil versus gemcitabine/docetaxel. Randomization may occur as early as vaccine is released (typically 3 - 4 weeks following tumor procurement) but no later than 8 weeks following tumor procurement. Randomization of patients will be stratified by Karnofsky Performance Status (KPS) ≥ 80% vs < 80%.

Patients will be managed in an outpatient setting. Hematologic function, liver enzymes, renal function and electrolytes will be monitored monthly. Blood for immune function analyses including IFNγ-ELISPOT analysis of cytotoxic T cell response to autologous tumor antigens will be collected at tissue procurement, baseline, and prior to product administration at Cycles 2, 4, end of treatment, and every 6 months thereafter.

Part 2 Methodology:

Based on the limited accrual to Part 1 of this study, Gradalis is opening Part 2 of this clinical protocol to assess the safety of Vigil immunotherapy in combination with irinotecan and temozolomide. Part 2 will be conducted at the same centers as Part 1, studying intradermal autologous Vigil cancer vaccine (1.0 x 10e7 cells/injection; minimum of 4 to a maximum of 12 administrations) in patients with metastatic Ewing's sarcoma Family of Tumors (ESFT) refractory or intolerant to at least 1 prior line of chemotherapy. Patients undergoing a standard surgical procedure (e.g., tumor biopsy or palliative resection) may have tumor tissue harvested for manufacture of investigational product. Patients meeting eligibility criteria including manufacture of a minimum of 4 immunotherapy doses of Vigil will be registered to receive: (i) oral temozolomide 100 mg/m2 daily (Days 1 - 5, total dose 500 mg/m2/cycle), (ii) irinotecan 50 mg/m2 daily (Days 1 - 5, total dose 250mg/m2/cycle), orally or irinotecan 20mg/m2 daily (Days 1 - 5, total dose 100mg/m2/cycle ), intravenously (iii) peg-filgrastim 100μg/kg (Day 6) subcutaneously (optional and may be administered at home), and (iv) Vigil 1.0 x 107 cells/injection, intradermally on Day 15 and every 3 weeks thereafter. One cycle = 21 days. Registration onto Part 2 may occur as early as one week but no later than 8 weeks following tumor procurement. Vigil is typically released approximately 3 weeks after the completion of the two-day manufacturing process.

Patients will be managed in an outpatient setting. Hematologic function, liver enzymes, renal function and electrolytes will be monitored. Blood for immune function analyses including IFNγ-ELISPOT analysis of cytotoxic T cell response to autologous tumor antigens will be collected at tissue procurement, post-procurement screening and prior to Day 15 Vigil administration at Cycles 2, 4, end of treatment, and every 6 months thereafter. Blood for ctDNA analysis will be collected prior to chemotherapy administration at baseline, Cycle 2 - Week 1 Day 1, Cycle 4 - Week 1 Day 1, and EOT.

ELIGIBILITY:
Tissue Procurement Inclusion Criteria:

Patients will be eligible for tissue procurement for the Vigil manufacturing process, if they meet all of the following criteria:

* Histologically confirmed Ewing's Sarcoma Family of Tumors (ESFT)
* Age ≥2 years
* Estimated survival ≥ 6 months
* Evidence of EWS translocation by FISH or RT-PCR or Next Generation Sequencing (NGS) Metastatic disease
* Refractory or intolerant to ≥ 2 lines of systemic chemotherapy (Part 1) or Refractory or intolerant to at least 1 line of systemic chemotherapy (Part 2)
* Planned standard of care surgical procedure (e.g., tumor biopsy or palliative resection or thoracentesis) and expected availability of a cumulative mass of ~10-30 grams tissue ("golf-ball" size) or pleural fluid estimated volume ≥ 500mL (must be primary tap) for immunotherapy manufacture
* Tumor intended for immunotherapy manufacture is not embedded in bone and does not contain luminal tissue (e.g., bowel, ureter, bile duct)
* Ability to understand and the willingness to sign a written informed consent document for tissue harvest

Tissue Procurement Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for tissue procurement for the Vigil manufacturing:

* Medical condition requiring any form of chronic systemic immunosuppressive therapy (steroid or other) except physiologic replacement doses of hydrocortisone or equivalent (no more than 30 mg hydrocortisone or 10 mg prednisone equivalent daily) for < 30 days duration
* Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected
* Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months
* Any documented history of autoimmune disease with exception of Type 1 diabetes on stable insulin regimen, hypothyroidism on stable dose of replacement thyroid medication, vitiligo, or asthma not requiring systemic steroids
* Known history of allergies or sensitivities to gentamicin
* Known hypersensitivity reactions to docetaxel or to other drugs formulated with polysorbate 80 that would preclude treatment with docetaxel (Part 1 only)
* History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.
* Known HIV or chronic Hepatitis B or C infection

Study Enrollment Inclusion Criteria:

Patients will be eligible for registration if they meet all of the following inclusion criteria:

* Successful manufacturing of at least 4 vials of Vigil
* Karnofsky performance status (KPS) ≥60% (Part 1) or KPS ≥80% (Part 2)
* Estimated survival ≥ 4 months (Part 1) or estimated survival of ≥6 months (Part 2)
* Normal organ and marrow function as defined below:

  * Absolute granulocyte count ≥1,500/mm3
  * Absolute lymphocyte count ≥400/mm3
  * Platelets ≥100,000/mm3
  * Total bilirubin ≤ institutional upper limit of normal
  * AST(SGOT)/ALT(SGPT) ≤2x institutional upper limit of normal
  * Creatinine <1.5 mg/dL
* Subject has recovered to CTCAE Grade 1 or better from all adverse events associated with prior therapy or surgery. Pre-existing motor or sensory neurologic pathology or symptoms must be recovered to CTCAE Grade 2 or better.
* If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry.
* Ability to understand and the willingness to sign a written informed protocol specific consent

Study Enrollment Exclusion Criteria:

Measureable disease is not a requirement for enrollment onto the trial.

In addition to the procurement exclusion criteria, patients will NOT be eligible for study registration and randomization if meeting any of the following criteria:

* Any anti-neoplastic therapy between tissue procurement for Vigil manufacture and start of study therapy
* Live vaccine used for the prevention of infectious disease administered < 30 days prior to the start of study therapy
* Post-surgery complication that in the opinion of the treating investigator would interfere with the patient's study participation or make it not in the best interest of the patient to participate

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Study Director — Gradalis, Inc.
Locations (6):
- United States (6):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Nicklaus Children's Hospital (Miami Children's Health System), Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - TOPA - Medical City Dallas Pediatric Hematology-Oncology, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghisoli M, Barve M, Schneider R, Mennel R, Lenarsky C, Wallraven G, Pappen BO, LaNoue J, Kumar P, Nemunaitis D, Roth A, Nemunaitis J, Whiting S, Senzer N, Fletcher FA, Nemunaitis J. Pilot Trial of FANG Immunotherapy in Ewing's Sarcoma. Mol Ther. 2015 Jun;23(6):1103-1109. doi: 10.1038/mt.2015.43. Epub 2015 Mar 19. PMID 25917459
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Ghisoli M, Barve M, Mennel R, Lenarsky C, Horvath S, Wallraven G, Pappen BO, Whiting S, Rao D, Senzer N, Nemunaitis J. Three-year Follow up of GMCSF/bi-shRNA(furin) DNA-transfected Autologous Tumor Immunotherapy (Vigil) in Metastatic Advanced Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1478-83. doi: 10.1038/mt.2016.86. Epub 2016 Apr 25. PMID 27109631
- [Background] Ghisoli M, Rutledge M, Stephens PJ, Mennel R, Barve M, Manley M, Oliai BR, Murphy KM, Manning L, Gutierrez B, Rangadass P, Walker A, Wang Z, Rao D, Adams N, Wallraven G, Senzer N, Nemunaitis J. Case Report: Immune-mediated Complete Response in a Patient With Recurrent Advanced Ewing Sarcoma (EWS) After Vigil Immunotherapy. J Pediatr Hematol Oncol. 2017 May;39(4):e183-e186. doi: 10.1097/MPH.0000000000000822. PMID 28338569

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Vigil Alone: Vigil immunotherapy 1.0 X 10^7 cells/injection; minimum of 4 to a maximum of 12 administrations every 28 days.
- Part 2: Vigil in Combination With Temozolomide and Irinotecan: (i) oral temozolomide 100 mg/m2 daily (Days 1 - 5, total dose 500 mg/m2/cycle), (ii) irinotecan 50 mg/m2 daily (Days 1 - 5, total dose 250mg/m2/cycle), orally or irinotecan 20mg/m2 daily (Days 1 - 5, total dose 100mg/m2/cycle ), intravenously (iii) peg-filgrastim 100μg/kg (Day 6) subcutaneously (optional and may be administered at home), and (iv) Vigil 1.0 x 107 cells/injection, intradermally on Day 15 and every 3 weeks thereafter. One cycle = 21 days.
Period: Overall Study
Arm/Group | Part 1: Vigil Alone | Part 1: Gemicitabine and Docetaxel | Part 2: Vigil in Combination With Temozolomide and Irinotecan
Started | 5 | 8 | 9
Completed | 5 | 7 | 9
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects registered to treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Vigil Alone | Part 1: Gemicitabine and Docetaxel | Part 2: Vigil in Combination With Temozolomide and Irinotecan | Total
Number analyzed (Participants) | 5 | 8 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 4 | 3 | 7
  Between 18 and 65 years | 5 | 4 | 6 | 15
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 4 | 13
  Male | 2 | 2 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 4 | 7 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 7 | 9 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Determined by Laboratory Assessments and Physical Examinations
Description: To determine safety profile of Vigil immunotherapy in combination with irinotecan and temozolomide with 30 days of last dose in patients with metastatic Ewing's sarcoma refractory or intolerant to at least 1 prior line of systemic chemotherapy.
  • To determine safety profile of Vigil immunotherapy in combination with irinotecan and temozolimidetemozolomide in patients with metastatic Ewing's sarcoma refractory or intolerant to at least 1 prior line of systemic chemotherapy.
Time Frame: 30 days of last treatment dosing
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Gemcitabine and Docetaxel: Gemcitabine 675 mg/m2 IV at 10 mg/m2/min D1 and Docetaxel 75 mg/m2 IV starting on D8 and given every 21 days.
Arm/Group | Part 1: Vigil Alone | Part 1: Gemcitabine and Docetaxel | Part 2: Vigil in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 5 | 8 | 9
Participants | 5 | 6 | 9

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) is defined as the time from randomization to the event of disease recurrence/progression defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) or death due to any cause. To determine the progression free survival of subjects dosed with Vigil immunotherapy in combination with irinotecan and temozolomide.
Time Frame: Estimated median 1.3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Vigil Alone | Part 1: Gemicitabine and Docetaxel | Part 2: Vigil in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 5 | 8 | 9
Participants | 5 | 6 | 9

3. Secondary Outcome: Overall Survival
Description: OS is defined as time from randomization to death or to the date of last follow-up. The date of last follow-up confirming survival will be used as the censoring date for subjects who are alive and/or do not have a known date of death.
Time Frame: Estimated median 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Vigil Alone | Part 1: Gemcitabine and Docetaxel | Part 2: Vigil in Combination With Temozolomide and Irinotecan
Number analyzed (Participants) | 5 | 8 | 9
Participants | 3 | 6 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for the duration of a patient's study treatment: from the first dose of the Investigational Product to 30 days following the last study treatment (up to 10 months).
Arm/Group | Part 1: Vigil Alone | Part 1: Gemicitabine and Docetaxel | Part 2: Vigil Plus Temozolomide and Irinotecan
All-Cause Mortality (participants affected / at risk) | 4/4 | 8/8 | 9/9
Serious Adverse Events (participants affected / at risk) | 2/5 | 5/8 | 5/9
Other Adverse Events (participants affected / at risk) | 2/5 | 5/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Vigil Alone (N=5) | Part 1: Gemicitabine and Docetaxel (N=8) | Part 2: Vigil Plus Temozolomide and Irinotecan (N=9)
Edema extremities (General disorders) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Brain mass (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Facial swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Platelets decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
WBC decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Vigil Alone (N=5) | Part 1: Gemicitabine and Docetaxel (N=8) | Part 2: Vigil Plus Temozolomide and Irinotecan (N=9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 6 (23)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (7) | 3 (16)
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Chronic heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Emesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (4) | 5 (12)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 6 (16)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Blood in stool (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (13)
Reflux esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Edema extremities (General disorders) | 2 (2) | 1 (2) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3) | 5 (13)
Fever (General disorders) | 1 (1) | 1 (2) | 3 (5)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0) | 2 (3)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral thrush (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes dermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelets decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
WBC decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Breath sounds decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 4 (7)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hip discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Jaw pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rib pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Swollen ankles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (4) | 1 (4)
Neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Foot drop (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Taste alteration (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blisters (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Facial swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Skin peeling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diaphoresis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pale skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
DVT (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to limited accrual to Part 1 of this study (rare disease), Gradalis opened Part 2 of this clinical protocol to assess the safety of Vigil immunotherapy in combination with irinotecan and temozolomide. Both parts of the study led to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-12): https://cdn.clinicaltrials.gov/large-docs/32/NCT02511132/Prot_SAP_000.pdf